CLINICAL TRIAL: NCT03230786
Title: A Double-blind, Placebo-controlled, Randomized Study to Evaluate the Efficacy and Safety of KBP-042 in Patients With Type 2 Diabetes
Brief Title: Study to Evaluate the Efficacy and Safety of KBP-042 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KeyBioscience AG (Industry)
Collaborators: Nordic Bioscience A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KBP042/CD/003; 2017-001061-24 (EudraCT Number)
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; KBP-042
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo QD for 12 weeks as add-on to metformin
  Interventions: Drug: Daily injection of KBP/placebo for 12 weeks as add-on to metformin
- 15µg KBP-042 QD (Experimental): Up to 15µg KBP-042 QD for 12 weeks as add-on to metformin
  Interventions: Drug: Daily injection of KBP/placebo for 12 weeks as add-on to metformin
- 30µg KBP-042 QD (Experimental): Up to 30µg KBP-042 QD for 12 weeks as add-on to metformin
  Interventions: Drug: Daily injection of KBP/placebo for 12 weeks as add-on to metformin
- 50µg KBP-042 QD (Experimental): Up to 50µg KBP-042 QD for 12 weeks as add-on to metformin
  Interventions: Drug: Daily injection of KBP/placebo for 12 weeks as add-on to metformin

INTERVENTIONS:
Drug: Daily injection of KBP/placebo for 12 weeks as add-on to metformin — Daily subcutaneous injection

SUMMARY:
This is a multicentre, randomized, double-blind, placebo-controlled, parallel-group Phase II trial of twelve weeks of KBP-042 administered as daily s.c. injections in subjects with Type 2 Diabetes Mellitus with inadequate glycaemic control while treated with a stable dose of metformin.

The trial is planned to be performed in Czech Republic, Denmark, Moldova, Poland, Romania and United Kingdom

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18-75 years of age, both inclusive, at the time of the first screening visit. Women must be either using adequate, highly effective methods of contraception, be post-menopausal or be considered sterile due to tubal ligation or other surgical procedures at the time of randomization. Sexually active men with a female partner of childbearing potential must agree in the use of highly effective method of contraception by the female partner throughout the trial period.
2. Subjects with type 2 diabetes mellitus diagnosis whose HbA1c levels are ≥7.0% and ≤10.0% (53 mmol/mol to 86 mmol/mol, respectively) at screening.
3. Stable therapy (for at least 90 days prior to randomization) with metformin.
4. Body mass index (BMI) ≥ 25.0 kg/m², and ≤ 45.0 kg/m².
5. The subject is able to understand and comply with protocol requirements.
6. The subject is able and willing to give written informed consent.

Exclusion Criteria:

1. Investigator considering the subject inappropriate for inclusion in the study based on medical interview and/or physical examination.
2. Past or present significant co-morbidity (other than type 2 diabetes mellitus) including, but not limited to: Active liver disease (other than asymptomatic non-alcoholic fatty liver disease), significant renal disease (including creatinine clearance < 45 ml/min by the Modification of Diet in Renal Disease (MDRD) method, congestive heart failure (NYHA class III or IV), myocardial infarction within the past 12 months, unstable angina pectoris.
3. Prior treatment in clinical trials with dual amylin and calcitonin receptor agonists (DACRAs).
4. Currently receiving medical treatment for obesity.
5. History of bariatric surgery.
6. Current alcohol abuse.
7. Current medical non-metformin anti-diabetic therapy, including SGLT2-inhibitors, DPP4-inhibitors (dipeptidyl peptidase 4 inhibitors), GLP-1 (Glucagon-like peptide 1) analogues, insulin and sulfonylureas, for a period of 90 days prior to randomization.
8. Use of thiazolidinediones (glitazones) lasting for more than one month within 90 days of randomization.
9. Regular use of insulin or insulin analogues.
10. History or presence of sensitivity or allergy to the study drug or drugs, to their components, or drugs of these classes or a history of drug or other allergy that contraindicates participation.
11. History of sarcoma or other malignancy within the past five years, except adequately treated basal cell or squamous cell carcinoma of the skin, or resected cervical atypia or carcinoma in situ.
12. Participation in a study trial with any investigational new drug (new chemical entity) within 90 days prior to the start of the study.
13. Pregnant females as determined by positive serum or urine human chorionic gonadotropin (hCG) test at screening or prior to randomization or during the treatment phase of the trial.
14. Breast-feeding women.
15. Known positive test results for hepatitis C antibodies, hepatitis B surface antigen, and HIV at screening.
16. ALT (alanine transaminase) or AST (aspartat transaminase) > 2.5 times the upper limit of normal at screening or other clinically significant liver function test abnormalities.
17. Clinically significant ECG abnormalities, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood HbA1c at 12 weeks versus placebo. | At 12 weeks

SECONDARY OUTCOMES:
Change from baseline in body weight at 12 weeks versus placebo. | At 12 weeks
Change from baseline in fasting serum glucose at 12 weeks versus placebo | At 12 weeks
Change from baseline in fasting serum insulin at 12 weeks versus placebo | At 12 weeks
Change from baseline in fasting serum glucagon at 12 weeks versus placebo | At 12 weeks
Proportion of subjects reaching a level of HbA1c below 7.0% (53 mmol/mol) at 12 weeks versus placebo | At 12 weeks

CONTACTS AND LOCATIONS:
Locations (30):
- Czechia (8):
  - Diabetologická a Obezitologická ambulance, České Budějovice
  - Vdoviak Miroslav MUDr. - Interní Ambulance, Karlovy Vary
  - Interní a Diabetologická ambulance, Clintrial s.r.o, Prague
  - Endokrinologicky Ústav, Prague
  - General University Hospital, Prague
  - Institute for Clinical and experimental Medicine, Prague
  - Diabet2 s.r.o, Prague
  - Interní a Diabetologická ambulance, Uherské Hradiště
- Denmark (7):
  - Bispebjerg Hospital, Endokrinologisk Afdeling, Bispebjerg, Copenhagen NV
  - Bioclinica, Ballerup Municipality, Copenhagen
  - Bioclinica, Aalborg, Jutland
  - Aarhus University Hospital, Endocrinlogy Department, Aarhus, Jutland
  - Sydvestjysk Sygehus, Esbjerg, Jutland
  - Bioclinica, Vejle, Jutland
  - Holbæk Sygehus, Holbæk
- Moldova (2):
  - Rtl Sm Srl/Scr, Chisinau
  - Rtl Sm Srl, Chisinau
- Poland (7):
  - Centrum Badań Klinicznych PI-House sp. z o.o., Gdansk
  - Specjalistyczna Praktyka Lekarska Piotr Kubalski, Grudziądz
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczno, Krakow
  - Prywatny Gabinet Lekarski i Wizyty Lekarskie Jan Ruxer, Lodz
  - Prywatny Gabinet Lekarski M. Horodecki (budynek Medicus), Opole
  - Centrum Medyczne Hygea, Tychy
  - Centrum Medyczne AMED, Warsaw
- Romania (5):
  - S.C. Policlinica CCBR S.R.L., Bucharest
  - Institutului Național de Diabet, Nutriție și Boli Metabolice "Prof.Dr. N.C. Paulescu", Bucharest
  - S.C Nicodiab S.R.L., Bucharest
  - S.C. Sfinx Medica S.R.L., Constanța
  - S.C. Mediab S.R.L., Târgu Mureş
- St. Pancras, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not to be shared